CLINICAL TRIAL: NCT05084937
Title: Celiac Disease in Childhood-Adulthood Transition (CeliCAT)
Brief Title: Celiac Disease in Childhood-Adulthood Transition
Acronym: CeliCAT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Kuopio University Hospital (Other); Turku University Hospital (Other Government); Seinajoki Central Hospital (Other); South Carelia Central Hospital (Other)
Responsible Party: Principal Investigator, Laura Kivelä, Principal Investigator, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R20068
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Celiac Disease; Celiac Disease in Children; Transition of Care; Follow-up; Diet, Gluten-Free
Keywords: celiac disease; adolescents; transition; follow-up; gluten-free diet; quality of life; health; symptoms
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Structured transition form is used with 50% of the study patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured transition (Active Comparator): With the help of CeliCAT form
  Interventions: Other: CeliCAT form
- Routine practices (No Intervention)

INTERVENTIONS:
Other: CeliCAT form — Systematic summary to support transition
  Arms: Structured transition

SUMMARY:
Aims of this study are to evaluate adolescents with celiac disease during their transition from pediatrics to adult care, and to develop better healthcare follow-up practices.

DETAILED DESCRIPTION:
Celiac disease is one of the most common chronic gastrointestinal diseases affecting 1-3% of population worldwide. It is treated with life-long and strict gluten-free diet. When dietary treatment is successful, prognosis of pediatric patients seems to be excellent whereas ongoing predisposition to gluten may increase the risk even to permanent complications. However, gluten-free diet may cause burden and restrictions in everyday life impairing quality of life. Regular follow-up is recommended to support the treatment and to detect early possible comorbidities and complications, but, in practice, patients are often lost to follow-up. Studies about the significance of follow-up and its optimal implementation are scarce. Pediatric patients form a special group here as they may not even remember the reason for the diagnosis if it was set in early childhood, and the education about the disease and its treatment are often given primarily to the caregivers. Responsibility of the treatment shifts to patients themselves in adolescence at the same time with other significant changes in life and they have more often challenges with gluten-free diet than other patients. Despite this, studies about the transition from pediatrics to adult-care are very few.

This study evaluates 13-19 years old patients diagnosed with celiac disease in childhood (<16 years of age) and compares them to adolescents without celiac disease in selected variables. Study focuses on healthcare follow-up practices and pilot a CeliCAT transition form in a randomized, controlled study design. The main hypothesis is that structured follow-up and transition of pediatric patients to adult care predicts better health, quality of life and adherence to the dietary treatment later in life. Data is collected with physical examination, questionnaires and with blood and urine samples. Follow-up is arranged at one and three years from the first visit.

ELIGIBILITY:
Inclusion Criteria:

* verified celiac disease diagnosis in childhood (<16 years of age)
* age 13-19 years at recruitment
* Finnish-speaking

Exclusion Criteria:

* disease or condition preventing the completing of the study questionnaire

Inclusion criteria for controls

* no celiac disease diagnosis
* age 13-19 years at recruitment
* Finnish-speaking

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to a gluten-free diet | At the onset of the study
  Assessed with questionnaire, celiac autoantibodies and urine GIP
Change in adherence to a gluten-free diet | After 1 and 3 years
  Assessed with questionnaire, celiac autoantibodies and urine GIP
Transition readiness | At the onset of the study
  Assessed with questionnaire
Change in transition readiness | After 1 and 3 years
  Assessed with questionnaire

SECONDARY OUTCOMES:
General health and health concerns | At the onset of the study
  Assessed with questionnaire
Change in general health and health concerns | After 1 and 3 years
  Assessed with questionnaire
Symptoms | At the onset of the study
  Assessed with questionnaire
Change in symptoms | After 1 and 3 years
  Assessed with questionnaire
Quality of life | At the onset of the study
  Assessed with questionnaire
Change in quality of life | After 1 and 3 years
  Assessed with questionnaire
Costs | At the onset of the study
  Assessed with questionnaire
Abnormalities in follow-up laboratory evaluations | At the onset of the study
  Assessed with blood sample
Abnormalities in physical examination | At the onset of the study
  Assessed with medical examination

CONTACTS AND LOCATIONS:
Locations (5):
- Finland (5):
  - Kuopio University Hospital, Kuopio
  - South Karelia Central Hospital, Lappeenranta
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere Celiac Disease Research Center, Tampere University, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No